CLINICAL TRIAL: NCT06188390
Title: Comparing Efficacy of Hydrodissection With Hyaluronic Acid vs 5% Dextrose for Carpal Tunnel Syndrome: A Randomized Controlled Trial and Ultrasonographic Evaluation of Median Nerve Gliding
Brief Title: Hydrodissection in Carpal Tunnel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TCRD-TPE-112-20(1/2)
Record Dates: First submitted 2023-08-17; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; hydrodissection; ultrasonography; median nerve gliding
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Hyaluronic acid and dextrose are both transparent, which is prepare by technician who is not participate in intervention and assessment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyaluronic acid group (Experimental): Hyaluronic acidwas injected under ultrasound guidance around wrist median nerve
  Interventions: Procedure: Ultrasound guided median nerve hydrodissection injection with Hyaluronic acid
- Dextrose group (Active Comparator): Dextrose was injected under ultrasound guidance around wrist median nerve
  Interventions: Procedure: Ultrasound guided median nerve hydrodissection injection with Dextrose water

INTERVENTIONS:
Procedure: Ultrasound guided median nerve hydrodissection injection with Hyaluronic acid — Hyaluronic acid was injected under ultrasound guidance around median nerve at the wrist
  Arms: Hyaluronic acid group
Procedure: Ultrasound guided median nerve hydrodissection injection with Dextrose water — Dextrose water was injected under ultrasound guidance around median nerve at the wrist
  Arms: Dextrose group

SUMMARY:
Compare the efficacy on carpal tunnel syndrome (CTS) treatment between hydrodissection with hyaluronic acid (HA) vs 5% dextrose

DETAILED DESCRIPTION:
Compare the efficacy on carpal tunnel syndrome treatment between hydrodissection with hyaluronic acid vs 5% dextrose through ultrasonographic evaluation.; 2) Evaluate the association of median nerve gliding results between using duplex Doppler ultrasound and B mode video with cross-correlation algorithm.

ELIGIBILITY:
Inclusion Criteria:

* 20-80 years old patients with carpal tunnel syndrome

Exclusion Criteria:

* pregnancy, Diabetes, hypothyroidism, uremia, rheumatoid arthritis, coagulopathy, cervical radiculopathy and patients who has ever received surgery for carpal tunnel syndrome or wrist fracture

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Boston CTS (carpal tunnel syndrome) questionnaire | before injection , 2 weeks, 3 months and 6 months after injection.
  The Boston CTS questionnaire is self-administered and is composed of two parts: the symptom severity scale (11 questions) and the functional status scale (8 questions).A final score is calculated for each scale (the sum of the individual scores divided by the number of items) and ranges from 1 to 5, with a higher score indicating a more severe handicap.

SECONDARY OUTCOMES:
Ultrasonography (B mode) of median nerve | before injection , 2 weeks, 3 months and 6 months after injection.
  Transverse ultrasonograms were obtained at the level of pisiform bone. Using electronic calipers, the CSA of the median nerve was measured by tracing the margin of the inner border of the perineural hyperechogenic rim that surrounded the hypoechoic median nerve , unit : mm2
Ultrasonography (duplex Doppler) of median nerve | before injection , 2 weeks, 3 months and 6 months after injection.
  An ultrasonography probe was placed longitudinally at the level of the lunate-capitate intercarpal joint to obtain a clear image of the median nerve. Longitudinal gliding excursions of the median nerve and flexor tendon were recorded using Doppler ultrasonography. The saved images were transferred to a personal coputer and analyzed by a researcher who was unaware of the individual and group identity of each image
Nerve conduction study (NCS) of median nerve | before injection , 3 months and 6 months after injection.
  Distal motor latencies of the median and ulnar nerve were respectively measured by placing a stimulating electrode at the wrist and a recording electrode 8 cm away from the stimulating electrode on the abductor pollicis brevis muscle and the adductor digiti minimi muscle. For sensory NCSs of the median and ulnar nerves, a standard distance of 14 cm was maintained between the stimulating electrode at the wrist and the recording electrodes at the ring finger on radial and ulnar sides

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Medicine and Rehabilitation, Taipei Tzu chi Hospital, Buddhist Tzu chi Medical Foundation, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lin MT, Liu IC, Syu WT, Kuo PL, Wu CH. Effect of Perineural Injection with Different Dextrose Volumes on Median Nerve Size, Elasticity and Mobility in Hands with Carpal Tunnel Syndrome. Diagnostics (Basel). 2021 May 9;11(5):849. doi: 10.3390/diagnostics11050849. PMID 34065073
- [Result] Su YC, Shen YP, Li TY, Ho TY, Chen LC, Wu YT. The Efficacy of Hyaluronic Acid for Carpal Tunnel Syndrome: A Randomized Double-Blind Clinical Trial. Pain Med. 2021 Nov 26;22(11):2676-2685. doi: 10.1093/pm/pnab109. PMID 33749798
- [Result] Babaei-Ghazani A, Moradnia S, Azar M, Forogh B, Ahadi T, Chaibakhsh S, Khodabandeh M, Eftekharsadat B. Ultrasound-guided 5% dextrose prolotherapy versus corticosteroid injection in carpal tunnel syndrome: a randomized, controlled clinical trial. Pain Manag. 2022 Sep;12(6):687-697. doi: 10.2217/pmt-2022-0018. Epub 2022 Jul 18. PMID 35848821